CLINICAL TRIAL: NCT05465473
Title: Effect of Low-level Laser Therapy During Maxillary Molar Distalization Using a Skeletally Anchored Appliance: A Prospective Clinical Study
Brief Title: Effect of Low-level Laser Therapy During Maxillary Molar Distalization Using a Skeletally Anchored Appliance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Talaat Hussein Ali, Assistant Lecturer, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 647/1760
Record Dates: First submitted 2022-07-08; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Class II Division 1 Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): will include 10 patients undergo distalization according to a standardized protocol
  Interventions: Other: Distalization
- Group II (Active Comparator): will include 10 patients undergo distalization assisted with low level laser therapy according to a standardized protocol
  Interventions: Other: Distalization

INTERVENTIONS:
Other: Distalization — Group I: will include 10 patients undergo distalization according to a standardized protocol. Group II: will include 10 patients undergo distalization assisted with low level laser therapy according to a standardized protocol.

SUMMARY:
study will be directed to evaluate the effect of low-level laser therapy during maxillary molar distalization using a skeletally anchored appliance

DETAILED DESCRIPTION:
Effect of low-level laser therapy during maxillary molar distalization using a skeletally anchored appliance

ELIGIBILITY:
Inclusion Criteria:

* 1- An age range from 14-17 years old. 2- All permanent teeth are present (except for third molars). 3- Bilateral dental Class II malocclusion. 4- Skeletal Class I or mild Class II relationship. 5- Normal or reduced vertical face height. 6- No posterior crowding or spaces.

Exclusion Criteria:

1. Patients who required surgery to correct skeletal discrepancies.
2. Patients with congenital dentoskeletal disorders.
3. Missed or mutilated teeth in maxillary arch.
4. Patients with poor oral hygiene and/or periodontally compromised patients.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2021-12-12 (Actual); Primary Completion 2022-08-12 (Estimated); Study Completion 2022-12-12 (Estimated)

PRIMARY OUTCOMES:
rate of molar distalization | from start of treatment until study completion, an average of 1 year
  rate of distalization of the maxillary first molars will be evaluated using direct clinical assessment and cast analysis according to standardized methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Al Azhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided